CLINICAL TRIAL: NCT06039917
Title: Effect of the Automatic Surveillance System on Surveillance Rate of Patients with Gastric Premalignant Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Shanghai Pudong Hospital (Other); The Eighth Hospital of Wuhan (Unknown); Jinjiang Municipal Hospital, Shanghai Sixth People's Hospital Fujian Campus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-AS2023-01
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Artificial Intelligence; Surveillance
Keywords: surveillance rate; automatic surveillance
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- With automatic surveillance system (Experimental): Patients were reminded of the surveillance time by an automatic surveillance system after the endoscopic and pathological results were available and before the surveillance time.
  Interventions: Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS)
- With manual reminder (Experimental): Patients were reminded of the surveillance time manually after the endoscopic and pathological results were available and before the surveillance time.
  Interventions: Other: Manually remind the patients
- Normal group (No Intervention): The patients in the control group were observed in the clinical natural state of surveillance without automatic surveillance system or manual reminder.

INTERVENTIONS:
Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) — An automatic surveillance (AS) system accurately identify patients with gastric premalignant lesions, assign surveillance intervals for different risks of patients and proactively follow up with patients at certain times.
  Arms: With automatic surveillance system
Other: Manually remind the patients — Medical staff remind patients to review manually.
  Arms: With manual reminder

SUMMARY:
In this study, we proposed a prospective study about the effect of the automatic surveillance system on surveillance rate of patients with gastric premalignant lesions. The enrolled patients were divided into group A with intelligent surveillance system, group B with manual reminder, and group C with natural state. The surveillance among the three groups will be compared.

DETAILED DESCRIPTION:
The adherence of doctors to published surveillance guidelines for patients with gastric premalignant lesions varies greatly, and surveillance of patients is critical but time-consuming. In previous studies we developed an automatic surveillance (AS) system to accurately identify patients with gastric premalignant lesions, assign surveillance intervals for different risks of patients and proactively follow up with patients in time. In this study, we proposed a prospective study about the effect of the automatic surveillance system on surveillance rate of patients with gastric premalignant lesions. The enrolled patients were divided into group A with intelligent surveillance system, group B with manual reminder, and group C with natural state. The surveillance among the three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older who undergo upper endoscopy.

Exclusion Criteria:

* 1)No contact information or invalid contact information.
* 2) The surveillance interval cannot be determined according to the surveillance guidelines, including no upper gastrointestinal pathology, therapeutic endoscopy or with history of previous gastrectomy, esophagectomy, or ESD, no dysplasia degrees, no biopsy sites, non-epithelial lesions, duodenal lesions, ulcer and so on.
* 3) Needless for surveillance or others.
* 4) High-grade intraepithelial neoplasia or cancer of the esophagus or stomach.
* 5) Low-grade intraepithelial neoplasia of the esophagus and Barrett's esophagus.
* 6) High-risk diseases or other special conditions for which the patient is deemed unsuitable for clinical trials by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
On-time Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with on-time surveillance, and the denominator is the number of all patients with gastric premalignant lesions requiring surveillance.

SECONDARY OUTCOMES:
Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance, and the denominator is the number of all patients with gastric premalignant lesions requiring surveillance.
Advance Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance in advance, and the denominator is the number of all patients with gastric premalignant lesions requiring surveillance.
Delayed Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with delayed surveillance, and the denominator is the number of all patients with gastric premalignant lesions requiring surveillance.
The accuracy of identifying patients with gastric premalignant lesions | 1 day At the time of enrollment
  The numerator is the number of patients correctly identified by automated surveillance system, and the denominator is the number of all enrolled patients with gastric premalignant lesions.
The accuracy of classifying risk levels | 1 day At the time of enrollment
  The numerator is the number of patients correctly classified by automated surveillance system, and the denominator is the number of all enrolled patients with gastric premalignant lesions.
The accuracy of assigning surveillance intervals | 1 day At the time of enrollment
  The numerator is the number of patients correctly assigned by automated surveillance system, and the denominator is the number of all enrolled patients with gastric premalignant lesions.
lesion progression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion progression, and the denominator is the number of all patients with gastric premalignant lesions undergoing surveillance.
lesion persistence rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion persistence, and the denominator is the number of all patients with gastric premalignant lesions undergoing surveillance.
lesion regression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion regression, and the denominator is the number of all patients with gastric premalignant lesions undergoing surveillance.
The incidence rate of early gastric cancer | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with early gastric cancer in surveillance endoscopy, and the denominator is the number of all patients with gastric premalignant lesions undergoing surveillance.
The incidence rate of gastric cancer | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with gastric cancer in surveillance endoscopy, and the denominator is the number of all patients with gastric premalignant lesions undergoing surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Yu, PhD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (4):
- China (4):
  - Jinjiang Municipal Hospital, Shanghai Sixth People's Hospital Fujian Campus, Quanzhou, Fujian
  - The Eighth Hospital of Wuhan, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No